CLINICAL TRIAL: NCT01615484
Title: Ex-vivo Perfusion and Ventilation of Lungs Recovered From Non-Heart-Beating Donors to Assess Transplant Suitability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Vitrolife (Industry); XVIVO Perfusion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNC-002 Vitrolife; 1UM1HL113115-01A1 (NIH)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-03

CONDITIONS: Emphysema; Chronic Obstructive Pulmonary Disease (COPD); Cystic Fibrosis; Pulmonary Fibrosis; Bronchiectasis; Sarcoidosis; Pulmonary Hypertension; Alpha-1 Antitrypsin Deficiency
Keywords: Lung Transplant; Emphysema; Chronic Obstructive Pulmonary Disease (COPD); Cystic Fibrosis; Pulmonary Fibrosis; Bronchiectasis; Sarcoidosis; Pulmonary Hypertension; Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis; Pulmonary Fibrosis; Bronchiectasis; Sarcoidosis; Hypertension, Pulmonary; alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ex-vivo lung perfusion (EVLP) with STEEN Solution™ (Experimental): The perfusion of the lungs will be performed using STEEN Solution™. The lungs will be physiologically assessed during ex vivo perfusion with STEEN Solution™ perfusate.
  Interventions: Procedure: Transplantation of lungs obtained from Non-Heart-Beating Donors (NHBDs) after ex-vivo perfusion w/ STEEN Solution™; Device: STEEN Solution™
- Lung transplant from conventional brain-dead organ donor (No Intervention): No experimental procedures will be carried out.

INTERVENTIONS:
Procedure: Transplantation of lungs obtained from Non-Heart-Beating Donors (NHBDs) after ex-vivo perfusion w/ STEEN Solution™ — After EVLP, lungs will be cooled in the circuit to room temperature, then flushed with cold Perfadex™, and taken to UNCH where they will have an ex-vivo CT scan. Lungs determined suitable will be offered to consented patients at UNC Hospitals and Duke University Medical Center based on Lung Allocation Score. Lungs not considered for transplantation may be subjected to different experiments but are not to be a part of this research study. In summary, lungs with good and stable function during EVLP will be transplanted into recipients as per current clinical practice.
  Arms: Ex-vivo lung perfusion (EVLP) with STEEN Solution™
Device: STEEN Solution™ — This solution is a buffered dextran and albumin-containing extracellular perfusate with an optimal colloid osmotic pressure developed specifically for extra-corporeal perfusion of lungs.
  Arms: Ex-vivo lung perfusion (EVLP) with STEEN Solution™

SUMMARY:
The purpose of this research study is to learn about the safety of transplanting lungs obtained from non-heart-beating donors (NHBDs) that have been ventilated (attached to a breathing machine or ventilator to deliver oxygen) and perfused with a lung perfusion solution (Steen solution™, made by Vitrolife). This ventilation and perfusion will be done outside the body (ex-vivo) in a modified cardiopulmonary bypass circuit (the kind of device used routinely during most heart surgeries). The purpose of performing ex-vivo perfusion and ventilation is to learn how well the lungs work, and whether they are likely safe to transplant.

ELIGIBILITY:
Inclusion Criteria:

* A recipient must meet the following requirement to enroll into the study:
* Requires a single or bilateral lung transplant and is listed for transplant at UNC or Duke
* Male or Female, 15 years of age or older.
* Subject or Subject's Representative provides a legally effective informed consent.
* Recipient does not have HIV, active Hepatitis or is colonized with Burkholderia cepacia.
* Potential subjects who have undergone previous lung transplants and meet all other inclusion criteria, are eligible for study participation.

Exclusion Criteria:

•Recipient fails to meet standard of care requirements for lung transplant, or decides not to participate.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. Egan, MD, MSc., Principal Investigator — UNC-Chapel Hill
Locations (2):
- United States (2):
  - UNC-Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Orens JB, Estenne M, Arcasoy S, Conte JV, Corris P, Egan JJ, Egan T, Keshavjee S, Knoop C, Kotloff R, Martinez FJ, Nathan S, Palmer S, Patterson A, Singer L, Snell G, Studer S, Vachiery JL, Glanville AR; Pulmonary Scientific Council of the International Society for Heart and Lung Transplantation. International guidelines for the selection of lung transplant candidates: 2006 update--a consensus report from the Pulmonary Scientific Council of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2006 Jul;25(7):745-55. doi: 10.1016/j.healun.2006.03.011. No abstract available. PMID 16818116
- [Background] Ingemansson R, Eyjolfsson A, Mared L, Pierre L, Algotsson L, Ekmehag B, Gustafsson R, Johnsson P, Koul B, Lindstedt S, Luhrs C, Sjoberg T, Steen S. Clinical transplantation of initially rejected donor lungs after reconditioning ex vivo. Ann Thorac Surg. 2009 Jan;87(1):255-60. doi: 10.1016/j.athoracsur.2008.09.049. PMID 19101308
- [Background] Mason DP, Thuita L, Alster JM, Murthy SC, Budev MM, Mehta AC, Pettersson GB, Blackstone EH. Should lung transplantation be performed using donation after cardiac death? The United States experience. J Thorac Cardiovasc Surg. 2008 Oct;136(4):1061-6. doi: 10.1016/j.jtcvs.2008.04.023. PMID 18954650
- [Background] Cypel M, Yeung JC, Hirayama S, Rubacha M, Fischer S, Anraku M, Sato M, Harwood S, Pierre A, Waddell TK, de Perrot M, Liu M, Keshavjee S. Technique for prolonged normothermic ex vivo lung perfusion. J Heart Lung Transplant. 2008 Dec;27(12):1319-25. doi: 10.1016/j.healun.2008.09.003. PMID 19059112
- [Background] Egan TM, Haithcock JA, Nicotra WA, Koukoulis G, Inokawa H, Sevala M, Molina PL, Funkhouser WK, Mattice BJ. Ex vivo evaluation of human lungs for transplant suitability. Ann Thorac Surg. 2006 Apr;81(4):1205-13. doi: 10.1016/j.athoracsur.2005.09.034. PMID 16564244
- [Background] Christie JD, Carby M, Bag R, Corris P, Hertz M, Weill D; ISHLT Working Group on Primary Lung Graft Dysfunction. Report of the ISHLT Working Group on Primary Lung Graft Dysfunction part II: definition. A consensus statement of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2005 Oct;24(10):1454-9. doi: 10.1016/j.healun.2004.11.049. Epub 2005 Jun 4. No abstract available. PMID 16210116
- [Background] Kim IK, Bedi DS, Denecke C, Ge X, Tullius SG. Impact of innate and adaptive immunity on rejection and tolerance. Transplantation. 2008 Oct 15;86(7):889-94. doi: 10.1097/TP.0b013e318186ac4a. PMID 18852649
- [Background] Moers C, Smits JM, Maathuis MH, Treckmann J, van Gelder F, Napieralski BP, van Kasterop-Kutz M, van der Heide JJ, Squifflet JP, van Heurn E, Kirste GR, Rahmel A, Leuvenink HG, Paul A, Pirenne J, Ploeg RJ. Machine perfusion or cold storage in deceased-donor kidney transplantation. N Engl J Med. 2009 Jan 1;360(1):7-19. doi: 10.1056/NEJMoa0802289. PMID 19118301
- [Background] Cypel M, Liu M, Rubacha M, Yeung JC, Hirayama S, Anraku M, Sato M, Medin J, Davidson BL, de Perrot M, Waddell TK, Slutsky AS, Keshavjee S. Functional repair of human donor lungs by IL-10 gene therapy. Sci Transl Med. 2009 Oct 28;1(4):4ra9. doi: 10.1126/scitranslmed.3000266. PMID 20368171
- [Background] Cypel M, Yeung JC, Liu M, Anraku M, Chen F, Karolak W, Sato M, Laratta J, Azad S, Madonik M, Chow CW, Chaparro C, Hutcheon M, Singer LG, Slutsky AS, Yasufuku K, de Perrot M, Pierre AF, Waddell TK, Keshavjee S. Normothermic ex vivo lung perfusion in clinical lung transplantation. N Engl J Med. 2011 Apr 14;364(15):1431-40. doi: 10.1056/NEJMoa1014597. PMID 21488765
- [Derived] Egan T, Blackwell J, Birchard K, Haithcock B, Long J, Gazda S, Casey N, Thys C. Assessment of Lungs for Transplant Recovered from Uncontrolled Donation after Circulatory Determination of Death Donors. Ann Am Thorac Soc. 2017 Sep;14(Supplement_3):S251. doi: 10.1513/AnnalsATS.201609-687MG. PMID 28945476

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Lungs were recovered from 35 NHBDs, 22 had EVLP. Two lung blocks were judged suitable, but not transplanted: No consented recipient available for #1, protocol time specifications could not be met for #2. As such, no subjects enrolled into EVLP arm.
Groups:
- Ex-vivo Lung Perfusion With STEEN Solution™: Transplantation of lungs obtained from Non-Heart-Beating Donors (NHBDs) after ex-vivo perfusion w/ STEEN Solution™ and CT scan.
Period: Overall Study
Arm/Group | Ex-vivo Lung Perfusion With STEEN Solution™ | Lung Transplant From Conventional Brain-dead Organ Donor
Started | 0 | 24
Completed | 0 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ex-vivo Lung Perfusion With STEEN Solution™ | Lung Transplant From Conventional Brain-dead Organ Donor | Total
Number analyzed (Participants) | 0 | 24 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 12 | 12
  >=65 years | 0 | 12 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 9 | 9
  Male | 0 | 15 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 0 | 20 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 24 | 24

OUTCOME MEASURES:

1. Primary Outcome: 30 Day Mortality and Graft Survival
Description: The primary objective evaluated for this study is recipient mortality and graft survival at 30 days post transplant. 30 day mortality and graft survival is used as a standard research assessment to evaluate post transplant outcomes.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Ex-vivo Lung Perfusion With STEEN Solution™ | Lung Transplant From Conventional Brain-dead Organ Donor
Number analyzed (Participants) | 0 | 24
Participants
  Alive | 0 | 22
  Deceased | 0 | 2

2. Primary Outcome: Primary Lung Graft Dysfunction (PGD)
Description: Primary Lung Graft Dysfunction (PGD) is an indicator for significant morbidity and mortality after lung transplantation.
  Grade 0: PaO2/FIO2 > 300 with normal chest radiograph; Grade 1: PaO2/FIO2 > 300 with diffuse infiltrates on the chest radiograph; Grade 2: PaO2/FIO2 between 200 and 300; Grade 3: PaO2/FIO2 < 200.
Time Frame: 24 and 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ex-vivo Lung Perfusion With STEEN Solution™ | Lung Transplant From Conventional Brain-dead Organ Donor
Number analyzed (Participants) | 0 | 24
Participants
  Grade 0 | 0 | 5
  Grade 1 | 0 | 9
  Grade 2 | 0 | 6
  Grade 3 | 0 | 4

3. Secondary Outcome: ICU Length of Stay
Description: The length of ICU stay in days is another standard research and clinical outcome assessment post transplant and has been selected as a secondary objective.
Time Frame: Time to Discharge, up to 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ex-vivo Lung Perfusion With STEEN Solution™ | Lung Transplant From Conventional Brain-dead Organ Donor
Number analyzed (Participants) | 0 | 24
Days |  | 6.91 (6.15)

4. Secondary Outcome: Day 7 Ventilator/ECMO Status
Description: Participants' status at Day 7 defined as the following: mechanical ventilation, extra-corporeal membrane oxygenator (ECMO), or extubated.
Time Frame: 7 Days Post Transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Ex-vivo Lung Perfusion With STEEN Solution™ | Lung Transplant From Conventional Brain-dead Organ Donor
Number analyzed (Participants) | 0 | 24
Participants
  Mechanical Ventilator |  | 4
  ECMO |  | 1
  Extubated |  | 19

5. Secondary Outcome: Recipient Mortality at 12 Months
Description: Recipient mortality at 12 months post transplant is being evaluated as a secondary objective.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ex-vivo Lung Perfusion With STEEN Solution™ | Lung Transplant From Conventional Brain-dead Organ Donor
Number analyzed (Participants) | 0 | 24
Participants
  Alive |  | 19
  Deceased |  | 5

6. Secondary Outcome: Bronchiolitis Obliterans Syndrome (BOS) Free Graft Survival
Description: Bronchiolitis Obliterans Syndrome (BOS) free graft survival at 12 months is being used as a secondary outcome.
Time Frame: 12 Months
Population: Excludes those who were deceased at Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Ex-vivo Lung Perfusion With STEEN Solution™ | Lung Transplant From Conventional Brain-dead Organ Donor
Number analyzed (Participants) | 0 | 19
Participants
  BOS-Free |  | 17
  BOS |  | 2

ADVERSE EVENTS:
Time Frame: From the date of transplant through 12 months post-op
Arm/Group | Ex-vivo Lung Perfusion With STEEN Solution™ | Lung Transplant From Conventional Brain-dead Organ Donor
All-Cause Mortality (participants affected / at risk) | 0/0 | 5/24
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/24
Other Adverse Events (participants affected / at risk) | 0/0 | 16/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ex-vivo Lung Perfusion With STEEN Solution™ (N=0) | Lung Transplant From Conventional Brain-dead Organ Donor (N=24)
Nausea and/or vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4)
Acute Rejection (Immune system disorders) | 0 (0) | 4 (4)
Pyrexia (Infections and infestations) | 0 (0) | 2 (2)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 6 (6)
Cytomegalovirus (CMV) (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)
Dehydration (General disorders) | 0 (0) | 2 (2)
Empyema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Lungs recovered from 35 NHBDs, 22 had EVLP. Two lung blocks judged suitable, but not transplanted: no consented recipient available for #1, protocol time specifications could not be met for #2. As such, no subjects enrolled into EVLP arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes